CLINICAL TRIAL: NCT07272629
Title: A Phase 1, Multicenter, Randomized, Double-blind, Double-dummy, Placebo- and Positive-controlled, 4-period Crossover Study to Evaluate the Effect of a Single Dose of Balinatunfib on Cardiac Repolarization in Healthy Adult Participants.
Brief Title: A Study to Evaluate the Effect of Single Oral Dose of Balinatunfib on Cardiac Repolarization in Healthy Adult Participants.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TES18591; U1111-1316-0289 (Other: WHO)
Record Dates: First submitted 2025-11-26; First posted 2025-12-09 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Cardiac Repolarization; Healthy Volunteers
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Williams design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Balinatunfib Treatment A (Experimental): Participants will receive a single oral dose of balinatunfib.
  Interventions: Drug: Balinatunfib; Drug: Placebo
- Balinatunfib Treatment B (Experimental): Participants will receive a single oral dose of balinatunfib.
  Interventions: Drug: Balinatunfib; Drug: Placebo
- Moxifloxacin Treatment C (Active Comparator): Participants will receive a single oral dose of moxifloxacin.
  Interventions: Drug: Moxifloxacin; Drug: Placebo
- Placebo Treatment D (Placebo Comparator): Participants will receive a single oral dose of balinatunfib matching placebo and moxifloxacin matching placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Balinatunfib — Pharmaceutical form: Tablet Route of administration: Oral
  Other Names: SAR441566
  Arms: Balinatunfib Treatment A; Balinatunfib Treatment B
Drug: Moxifloxacin — Pharmaceutical form: Tablet Route of administration: Oral
  Arms: Moxifloxacin Treatment C
Drug: Placebo — Pharmaceutical form: Tablet Route of administration: Oral

SUMMARY:
This is a Phase 1, multicenter, randomized, double-blind, double-dummy, single dose, placebo- and positive-controlled, 4-sequence, 4-treatment, 4-period crossover study.

ELIGIBILITY:
Inclusion Criteria:

* Age: Healthy males and/or females aged 18 to 55 (inclusive) at consent signing.
* Certified healthy based on history, physical exam, vitals, ECG, and labs with no abnormalities.
* Weight: 50-100 kg (male), 40-90 kg (female); BMI 18-30 kg/m² inclusive.
* Sex-based eligibility: All males must use effective contraception or remain abstinent and avoid sperm donation for 3 months post-dose. Females must use highly effective contraception, not be pregnant or breastfeeding, and test negative for pregnancy before treatment.

Exclusion Criteria:

* History of significant systemic diseases (hematologic, renal, endocrine, pulmonary, GI, cardiac, hepatic, psychiatric, neurologic, infectious, allergic; except mild seasonal allergies).
* Clinically significant ECG abnormalities.
* Frequent headaches or migraines, and recurrent nausea or vomiting (over twice monthly).
* Blood donation within 2 months.
* Symptomatic or significant postural hypotension.
* Drug hypersensitivity or significant allergies, including to study drugs.
* History of drug/alcohol abuse.
* Tobacco use within 3 months prior to Day 1.
* History of Hepatitis B/C, TB, or invasive opportunistic infections.
* Malignancy within 5 years (except treated non-metastatic skin cancer).
* Adverse reaction to balinatunfib, moxifloxacin, or quinolones.
* Any medication (except hormonal contraception/HRT) within 14 days or 5× half-life.
* Biologics within 4 months prior.
* Vaccines: non-live within 4 weeks, live within 3 months before or during study.
* Current or recent participation in another interventional study within 30 days.
* Positive for HBsAg, anti-HBc, anti-HCV, anti-HIV1/2.
* Positive urine drug screen.
* Positive alcohol breath test.
* Positive urine cotinine test.
* History of long QT syndrome.
* Risk factors for TdP.
* Moxifloxacin contraindications.
* Low potassium (<3.5 mmol/L).
* Low magnesium (<0.7 mmol/L).

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Both males and females aged 18-55 years are eligible, with at least 30% representation from each gender.
Enrollment: 44 (Estimated)
Dates: Start 2025-12-04 (Actual); Primary Completion 2026-04-27 (Estimated); Study Completion 2026-04-27 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the QT interval corrected using the Fridericia formula (QTcF) centrally assessed using a semi-automatic reading | Baseline to day 2

SECONDARY OUTCOMES:
Change from baseline in heart rate (HR) | Day 1 to Day 2
Change from baseline in QT interval | Baseline to day 2 of each period
Change from baseline in QT interval corrected using the Bazett formula (QTcB) | Baseline to day 2 of each period
Change from baseline in population specific QT correction (QTcN) interval | Baseline to day 2 of each period
Change from baseline in QRS interval | Baseline to day 2 of each period
Change from baseline in PR interval | Baseline to day 2 of each period
Safety for electrocardiogram (ECG) parameters | Baseline to day 83
Maximum plasma concentration (Cmax) for balinatunfib | Baseline to day 6 of each period
Time to reach the maximum concentration (tmax) for balinatunfib | Baseline to day 6 of each period
Area under the curve (AUC) for balinatunfib | Baseline to day 6 of each period
Maximum plasma concentration (Cmax) for balinatunfib metabolite M8 | Baseline to day 6 of each period
Time to reach the maximum concentration (tmax) for balinatunfib metabolite M8 | Baseline to day 6 of each period
Area under the curve (AUC) for balinatunfib metabolite M8 | Baseline to day 6 of each period
Number of participants experiencing treatment-emergent adverse events (TEAEs) including adverse events of special interest (AESIs) and serious adverse events (SAEs) | Baseline to Day 83
Number of participants with clinical laboratory and vital signs abnormalities (potentially clinically significant abnormality) | Baseline to Day 83

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - FORTREA CLINICAL RESEARCH UNIT INC- Site Number : 8400002, Dallas, Texas
  - FORTREA CLINICAL RESEARCH UNIT INC- Site Number : 8400001, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: TES18591 Plain Language Results Summary — https://sanofi.trialsummaries.com/Study/StudyDetails?id=26955&tenant=MT_SNY_9011